CLINICAL TRIAL: NCT02130609
Title: Skintel Integration Study for Use With the Elite+ Laser System
Brief Title: Skintel Integration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN13-SkinTel-Elite+-01
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Skin Type From I-VI on Non-hair Bearing Skin

STUDY DESIGN:
Intervention Model Description: Even though this study has recruited more than 10 participants, it is a feasibility study, designed to test the prototype rather than measuring health outcomes. It is to confirm the operating specifications before beginning a full clinical trial. The objective of this study is to improve the treatment guidelines for the Elite+ by determining the maximum safe settings for skin and correlate them to measurement of Melanin Index (MI).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skintel (Experimental)
  Interventions: Device: Skintel

INTERVENTIONS:
Device: Skintel

SUMMARY:
The objective of this study is to improve the treatment guidelines for the Elite+ by determining the maximum safe settings for skin and correlate them to measurement of Melanin Index (MI) (MI).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to read, understand, and sign the Informed Consent Form
* Willing and able to comply with all study requirements

Exclusion Criteria:

* Hypersensitivity to light in the near infrared wavelength region
* Sun-damaged skin (treatment contraindicated with Alex laser only)
* Unprotected sun exposure (for Alex laser within four weeks of treatment; for
* Nd:YAG laser within one week of treatment), including the use of tanning beds or
* tanning products, such as creams, lotions and sprays
* Take medication which is known to increase sensitivity to sunlight
* Seizure disorders triggered by light
* Take anticoagulants
* Take or have taken oral isotretinoin, such as Accutane®, within the last six months
* Take medication that alters the wound-healing response
* History of healing problems or history of keloid formation
* Active localized or systemic infection, or an open wound in area being treated
* Significant systemic illness or an illness localized in area being treated
* History of skin cancer or suspicious lesions
* Lupus
* Have received or are receiving or gold therapy
* Pregnancy, planning on becoming pregnant or have been pregnant recently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
improve the treatment guidelines for the Elite+ by determining the maximum safe settings for skin and correlate them to measurement of Melanin Index | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean Doherty, MD, Principal Investigator